CLINICAL TRIAL: NCT03928184
Title: A Phase 3, 56-Week, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Utilizing Patient-Reported and Radiographic Outcomes to Evaluate the Efficacy and Safety of a Single Injection of SM04690 Injected in the Target Knee Joint of Moderately to Severely Symptomatic Osteoarthritis Subjects
Brief Title: A Study Utilizing Patient-Reported and Radiographic Outcomes and Evaluating the Safety and Efficacy of Lorecivivint (SM04690) for the Treatment of Moderately to Severely Symptomatic Knee Osteoarthritis
Acronym: STRIDES-X-ray
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SM04690-OA-11
Record Dates: First submitted 2019-04-23; First posted 2019-04-26 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Knee Osteoarthritis
Keywords: SM04690; Wnt pathway inhibitor; osteoarthritis; Samumed; lorecivivint
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — lorecivivint

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 0.07 mg lorecivivint (Experimental): One intra-articular injection of 0.07 mg lorecivivint in 2 ml vehicle
  Interventions: Drug: Lorecivivint
- Vehicle (Placebo Comparator): One intra-articular injection of 0 mg lorecivivint in 2 ml vehicle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lorecivivint — Healthcare professional-administered intra-articular injection; performed on Day 1
  Other Names: SM04690
  Arms: 0.07 mg lorecivivint
Drug: Placebo — Healthcare professional-administered intra-articular injection; performed on Day 1
  Arms: Vehicle

SUMMARY:
This phase 3 study is a multicenter, randomized, double-blind, placebo-controlled study of lorecivivint injected intra-articularly (IA) into the target knee (most painful) joint of moderately to severely symptomatic osteoarthritis (OA) subjects at a single dose of 0.07 mg lorecivivint per 2 mL injection. This study will utilize radiographs and patient reported outcomes (PROs) to evaluate the safety and efficacy of lorecivivint.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 40 and 80 years of age, inclusive, in general good health apart from their knee OA
2. Ambulatory (single assistive devices such as canes allowed if needed less than 50% of the time, subjects requiring a walker are excluded)
3. Diagnosis of femorotibial OA in the target knee by standard American College of Rheumatology (ACR) criteria at the Screening Visit (clinical AND radiographic criteria); OA of the knee is not to be secondary to any rheumatologic conditions (e.g., rheumatoid arthritis)
4. mJSW by radiograph between 1.5 and 4 mm, inclusive, in the target knee within 12 weeks of the Screening Visit as assessed by independent central readers
5. Radiographic disease Stage 2 or 3 in the target knee within 12 weeks of the Screening Visit according to the Kellgren-Lawrence (KL) grading of knee OA as assessed by independent central readers
6. Pain compatible with OA of the knee(s) for at least 26 weeks prior to the Screening Visit
7. Primary source of pain throughout the body is due to OA in the target knee
8. Body mass index (BMI) ≤ 40 kg/m2 at the Screening Visit
9. Widespread Pain Index (WPI) score of ≤ 4 and a Symptom Severity Question 2 (SSQ2) score of ≤ 2 at the Screening Visit and Day 1
10. Pain NRS scores recorded for the target knee on at least 4 out of the 7 days immediately preceding Day 1
11. Pain NRS scores recorded for the nontarget knee on at least 4 out of the 7 days immediately preceding Day 1
12. Daily OA knee pain diary average NRS intensity score ≥ 4 and ≤ 8 in the target knee on the 11-point (0-10) NRS scale for the 7 days immediately preceding Day 1
13. Daily OA knee pain diary average NRS intensity score < 4 in the nontarget knee on the 11-point (0-10) NRS scale for the 7 days immediately preceding Day 1
14. WOMAC Pain of 20-40 (out of 50) for the target knee at baseline regardless of if the subject is on symptomatic oral treatment (baseline questionnaire completed during the screening period prior to randomization)
15. WOMAC Function of 68-136 (out of 170) for the target knee at baseline regardless of if the subject is on symptomatic oral treatment (baseline questionnaire completed during the screening period prior to randomization)
16. Willingness to use an electronic diary daily in the evening for the screening period and 56-week study duration
17. Negative drug test for amphetamine, buprenorphine, cocaine, methadone, opiates, phencyclidine (PCP), propoxyphene, barbiturates, benzodiazepine, methaqualone, and tricyclic antidepressants, unless any of these drugs are allowed per protocol and prescribed by a physician to treat a specific condition
18. Subjects with depression or anxiety must be clinically stable for at least 12 weeks prior to the Screening Visit and, if on treatment for depression or anxiety, be on at least 12 weeks of stable therapy
19. Full understanding of the requirements of the study and willingness to comply with all study visits and assessments
20. Subjects must have read and understood the informed consent form (ICF), and must have signed and dated it prior to any study-related procedure being performed

Exclusion Criteria:

1. Pregnant women, breastfeeding woman, and women who are not post-menopausal (defined as 12 months with no menses without an alternative medical cause) or permanently surgically sterile (includes hysterectomy, bilateral salpingectomy, and bilateral oophorectomy), who have a positive or indeterminate pregnancy test result at the Screening Visit or Day 1
2. Women who are not post-menopausal or permanently surgically sterile who are sexually active, and who are not willing to use birth control during the study period
3. Men who are sexually active and of reproductive potential, who have partners who are capable of becoming pregnant, and who are not willing to use birth control during the study period
4. Significant malalignment of anatomical axis (medial angle formed by the femur and tibia) of the target knee (varus > 10°, valgus > 10°) by radiograph within 12 weeks of the Screening Visit as assessed by independent central readers
5. Partial or complete joint replacement in either knee
6. Currently requires use of a lower extremity prosthesis, and/or a structural knee brace (i.e., a knee brace that contains hardware)
7. Any surgery (e.g., arthroscopy) in either knee within 26 weeks prior to Day 1
8. Intra-articular (IA) injection into the target knee with a therapeutic aim including, but not limited to, hyaluronic acid, platelet-rich plasma (PRP),and stem cell therapies within 26 weeks prior to Day 1, or IA glucocorticoids within 12 weeks prior to Day 1
9. Effusion of the target knee clinically requiring aspiration within 12 weeks prior to Day 1
10. Use of electrotherapy, acupuncture, physical therapy, therapeutic ultrasound, and/or chiropractic treatments for knee OA within 4 weeks prior to Day 1
11. Any bone fracture(s) within 26 weeks prior to the Screening Visit
12. Previous treatment with SM04690
13. Subjects who have previously failed screening on this protocol and fail to meet rescreening criteria
14. Participation in a clinical research trial that included the receipt of an investigational product (IP) or any experimental therapeutic procedure within 26 weeks prior to the Screening Visit, or planned participation in any such trial
15. Treatment with systemic (oral, intramuscular, or intravenous) glucocorticoids ≥10 mg prednisone or the equivalent per day within 4 weeks prior to Day 1, or subjects on <10 mg prednisone or the equivalent per day who have not maintained a stable regimen for at least 2 weeks prior to Day 1 in the opinion of the Investigator
16. Use of centrally acting analgesics within 12 weeks prior to Day 1
17. Use of anticonvulsants within 12 weeks prior to Day 1
18. Subjects requiring the use of opioids > 1x per week within 12 weeks prior to Day 1
19. Topical local anesthetic agents (gels, creams, or patches such as the Lidoderm patch) used for the treatment of knee OA within 7 days of Day 1
20. Planned surgery scheduled during the study period, not including non-surgical invasive procedures conducted for a diagnostic or therapeutic purpose scheduled during the study period
21. History of malignancy within the last 5 years, not including subjects with prior history of adequately treated in situ cervical cancer or basal or squamous cell skin cancer
22. Clinically significant abnormal screening hematology values, blood chemistry values, or urinalysis values as determined by the Investigator
23. Any condition, that, in the opinion of the Investigator, constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation
24. Other conditions that, in the opinion of the Investigator, could affect study endpoint assessments of either knee, including, but not limited to, peripheral neuropathy (e.g., diabetic neuropathy), symptomatic hip osteoarthritis, symptomatic degenerative disc disease, and patellofemoral syndrome
25. Comorbid conditions that could affect study endpoint assessments of the target knee, including, but not limited to, rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus, gout or pseudogout, and fibromyalgia
26. History of mania, bipolar disorder, psychotic disorder, schizophrenia, or schizoaffective disorder
27. Any known active infections, including urinary tract infection, upper respiratory tract infection, sinusitis, suspicion of IA infection, hepatitis B or hepatitis C infection, and/or infections that may compromise the immune system such as human immunodeficiency virus (HIV) at Day 1
28. Any chronic condition that has not been well controlled or subjects with a chronic condition who have not maintained a stable therapeutic regimen of a prescription therapy in the opinion of the Investigator.
29. Hemoglobin A1c (HbA1c) >9 at the Screening Visit
30. If using NSAIDs and/or acetaminophen, subjects who have not maintained a stable regimen in the opinion of the Investigator for at least 4 weeks prior to Day 1
31. Any contraindications for an IA injection in the target knee in the opinion of the Investigator
32. Subjects who have a current or pending disability claim, workers' compensation, or litigation(s) that may compromise response to treatment
33. Subjects who are immediate family members (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with the study at any investigative site, or are directly affiliated with the study at any investigative site
34. Subjects employed by Samumed, LLC, or any of its affiliates or development partners (that is, an employee, temporary contract worker, or designee) responsible for the conduct of the study, or who are immediate family members (spouse, parent, child, or sibling; biological or legally adopted) of said employees responsible for the conduct of the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in OA pain in the target knee (pain NRS) | Baseline and Week 12
  Evaluate change from baseline OA pain in the target knee as assessed by the weekly averages of daily pain numeric rating scale (NRS). The pain NRS is an 11-point scale [0-10] for subject self-reporting of average knee pain in the last 24 hours; 0 indicates no pain, and 10 represents the worst possible pain.

SECONDARY OUTCOMES:
Change from baseline in OA pain in the target knee (Pain NRS) | Baseline, Weeks 24 and 52
  Evaluate change from baseline OA pain in the target knee as assessed by the weekly averages of daily pain Numeric Rating Scale (NRS). The pain NRS is an 11-point scale [0-10] for subject self-reporting of average knee pain in the last 24 hours; 0 indicates no pain, and 10 represents the worst possible pain.
Change from baseline in OA function in the target knee (WOMAC Function) | Baseline, Weeks 12, 24 and 52
  Evaluate change from baseline OA function in the target knee as assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) physical function subscore (WOMAC Function). The WOMAC is a widely-used, proprietary outcome measurement tool used to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions), and physical functioning (17 questions) of the joints. Each question is measured on a scale from 0 (lowest pain/lowest stiffness/highest function) to 4 (highest pain/highest stiffness/lowest function). The WOMAC Function subscore ranges from 0 to 68.
Change from baseline in OA disease activity (Patient Global Assessment) | Baseline, Weeks 12, 24 and 52
  Evaluate change from baseline OA disease activity as assessed by Patient Global Assessment. The Patient Global Assessment is an 11-point [0-10] Numeric Rating Scale [NRS] on which the subjects will rate how they feel their target knee OA is doing, considering all the ways in which their target knee OA may affect them. The NRS is anchored by descriptors at each end ("Very Good" on the left and "Very Bad" on the right).
Change from baseline in usage of nonsteroidal anti-inflammatory drugs (NSAIDs) and acetaminophen for target knee OA pain | Baseline and Week 52

OTHER OUTCOMES:
Change from baseline in serum bone biomarkers | Baseline and Week 56
  Evaluate change from baseline in serum bone biomarkers N-terminal propeptides of procollagen type I [PINP] and β-C-terminal telopeptide [β-CTX]
Change from baseline in a serum cartilage biomarker | Baseline and Week 56
  Evaluate change from baseline in serum cartilage biomarker cartilage oligomeric matrix protein [COMP]
Change from baseline in medial joint space width (mJSW) in the target knee | Baseline and Week 52
  Evaluate change from baseline in mJSW as documented by radiograph of the target knee
Change from baseline in health-related quality of life (HRQOL) | Baseline and Week 52
  Evaluate change from baseline in HRQOL as assessed by the 36-Item Short Form Health Survey (SF-36). The SF-36 consists of eight scaled scores which are the weighted sums of the questions in their section (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health). Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. A score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change from baseline in OA pain in the target knee (WOMAC Pain) | Baseline, Weeks 12, 24 and 52
  Evaluate change from baseline in OA pain in the target knee as assessed by WOMAC pain subscore (WOMAC Pain). The WOMAC is a widely-used, proprietary outcome measurement tool used to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions), and physical functioning (17 questions) of the joints. Each question is measured on a scale from 0 (lowest pain/lowest stiffness/highest function) to 4 (highest pain/highest stiffness/lowest function). The WOMAC Pain subscore ranges from 0 to 20.
Change from baseline in OA pain, function and stiffness (WOMAC Total score) | Baseline, Weeks 12, 24 and 52
  Evaluate change from baseline in OA pain, function and stiffness as a composite outcome measure as assessed by WOMAC Total score. The WOMAC is a widely-used, proprietary outcome measurement tool used to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions), and physical functioning (17 questions) of the joints. Each question is measured on a scale from 0 (lowest pain/lowest stiffness/highest function) to 4 (highest pain/highest stiffness/lowest function). WOMAC Total is a composite of the three domains (pain/stiffness/function) with a total score of 0 to 96.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Yazici, M.D., Study Director — Biosplice Therapeutics, Inc.
Locations (91):
- United States (91):
  - Research Site, Birmingham, Alabama
  - Research Site, Peoria, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Garden Grove, California
  - Research Site, Norco, California
  - Research Site, Pomona, California
  - Research Site, San Diego, California
  - Research Site, San Marcos, California
  - Research Site, Spring Valley, California
  - Research Site, Westminster, California
  - Research Site, Boulder, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Waterbury, Connecticut
  - Research Site, Clearwater, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Orlando, Florida
  - Research Site, Oviedo, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Sunrise, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Winter Haven, Florida
  - Research Site #1, Winter Park, Florida
  - Research Site #2, Winter Park, Florida
  - Research Site, Marietta, Georgia
  - Research Site, Newnan, Georgia
  - Research Site, Stockbridge, Georgia
  - Research Site, Woodstock, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Meridian, Idaho
  - Research Site, Bloomington, Illinois
  - Research Site, Gurnee, Illinois
  - Research Site, Oak Brook, Illinois
  - Research Site, Rockford, Illinois
  - Research Site, Anderson, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Kansas City, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Monroe, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Wheaton, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Bay City, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Hazelwood, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, La Vista, Nebraska
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Albuquerque, New Mexico
  - Research Site, Great Neck, New York
  - Research Site, Hartsdale, New York
  - Research Site, New York, New York
  - Research Site 1, New York, New York
  - Research Site 2, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Williamsville, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Leland, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Fort Mill, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Austin, Texas
  - Research Site, Bedford, Texas
  - Research Site, Carrollton, Texas
  - Research Site, Dallas, Texas
  - Research Site, Edinburg, Texas
  - Research Site, Houston, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Draper, Utah
  - Research Site, Murray, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tambiah J, Kennedy S, Swearingen C, McAlindon T, Yazici Y. Impact of structural severity on outcomes in knee osteoarthritis: an analysis of data from phase 2 and phase 3 lorecivivint clinical trials. Rheumatology (Oxford). 2025 May 1;64(5):2583-2590. doi: 10.1093/rheumatology/keae610. PMID 39495154